CLINICAL TRIAL: NCT07250919
Title: Donor and Recipient Mismatch in Liver Transplantation - Time for Reconsideration?
Brief Title: Donor and Recipient Mismatch in Liver Transplantation
Acronym: DR-MM in LT
Status: Completed | Type: Observational
Sponsor: University of Jena (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Nicola Sariye Pollmann, Principal Investigator, University of Jena
Other Study IDs: 20-5877.4
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-10

CONDITIONS: Patient Survival; Graft Survival; Liver Disease (Alcoholic or Not); Liver Transplant Surgery
Keywords: liver transplantation; patient survival; gender mismatch; long-term outcome; organ allocation
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GM +: Liver transplant recipients with gender mismatch
- GM -: Liver transplant recipients without gender mismatch

SUMMARY:
This observational study aims to investigate the impact of gender disparity between donors and recipients on long-term outcomes after liver transplantation (LT). The study aims to answer the following question:

Does gender mismatch lower the possibility of survival after liver transplantation? Participants demonstrate gender dicrepancies between donors and recipients as regular concept in LT. The retrospective cohort study investigates the impact over a long-term follow up of 10 years.

DETAILED DESCRIPTION:
The study involves patients who undergo liver transplantation at the Ajmera Transplant Centre Toronto from 2014 until 2022. The observation period ended at the first January 2025 to provide a minimal follow up of 24 months.

Liver transplant recipients with gender mismatch (A) will be compared with liver transplant recipients without gender mismatch (B).

Liver transplantation is the only curative treatment for people with end stage liver disease. Gender mismatch between donor and recipient, particularly, the combination of a female donor to male recipient has been controversial in the past. Identifying risk factors that could affect the survival of the graft and recipient is of the utmost importance.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18

Exclusion Criteria:

* Cases of retransplantation
* Combined organ transplantation
* Cases with >30% of missing values

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since gender discrepancies are studied, the participant are identified by their biological gender, including male and female.
Study Population: Patients who underwent liver transplantation at who at the Ajmera transplant centre, Toronto between 2014 and 2022
Sampling Method: Probability Sample
Enrollment: 1146 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Patient survival | Liver transplantation between 01.01.2014 and 01.01.2022, Patient Survival: observatory period between 01.01.2014 and 01.01.2024
  Overall survival of patients who underwent liver transplantation at the Ajmera transplant centre toronto between 2014 and 2022

CONTACTS AND LOCATIONS:
Locations (1):
- Ajmera Transplant Centre, Toronto General Hospital, University Health Network, Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
The investigators consider not to share IPD before publishing the study.

REFERENCES:
- [Background] Ghinolfi D, Melandro F, Torri F, Martinelli C, Cappello V, Babboni S, Silvestrini B, De Simone P, Basta G, Del Turco S. Extended criteria grafts and emerging therapeutics strategy in liver transplantation. The unstable balance between damage and repair. Transplant Rev (Orlando). 2021 Dec;35(4):100639. doi: 10.1016/j.trre.2021.100639. Epub 2021 Jul 16. PMID 34303259

DOCUMENTS (1):
  • Study Protocol (2025-11-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT07250919/Prot_001.pdf